CLINICAL TRIAL: NCT04793282
Title: The Benefits of Telephone Follow-Up After a Mental Health Assessment in an Emergency Department
Brief Title: The Benefits of Telephone Follow-up (TFU)
Acronym: TFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brandon University (Other)
Responsible Party: Principal Investigator, Alana Prejet, Principal Investigator, Brandon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BrandonU
Record Dates: First submitted 2021-02-23; First posted 2021-03-11 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Mental Health Issue
Keywords: Telephone follow up

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Post-test satisfaction
  Interventions: Behavioral: Telephone Follow-up
- Experimental (Experimental): Treatment and satisfaction
  Interventions: Behavioral: Telephone Follow-up

INTERVENTIONS:
Behavioral: Telephone Follow-up — Telephone Follow-up within 72 hours to discuss psycho education, discharge planning and clarify any questions they may have.

SUMMARY:
This study will investigate the impact of a brief telephone follow-up following a mental health assessment in the emergency department. The purpose of the telephone call will be to provide psycho-education, clarify any questions and reinforce discharge planning.

DETAILED DESCRIPTION:
This is a randomized controlled trial. The experimental group will receive a phone call within 72 hours of discharge to provide psycho education, clarify any questions they may have and to reinforce discharge plans made in the ED. The control group will not receive this phone call. Within 30 days of discharge, both groups will receive a phone call to collect data on treatment compliance including medication and follow-up adherence and if any additional visits to the Emergency Department were necessary.

ELIGIBILITY:
Inclusion Criteria

* Discharged from the ED
* Age of majority
* Competent.

Exclusion Criteria

* Incompetent,
* Under 18
* Admitted to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Emergency Department readmission rates | 30 days.
  Does a telephone call reduce readmission rates?

SECONDARY OUTCOMES:
Satisfaction with care in the Emergency Department using a 7 point Likert Scale as a function of the telephone follow up. | 30 days.
  Various measures of satisfaction in care provided in Emergency Department. Higher scores indicate higher satisfaction.
Adherence to pharmacological interventions and follow-up appointments. | 30 days.
  Adhering to pharmacological interventions and follow-up appointments by self rating on a 7 point Likert Scale. Higher scores indicate greater adherence to treatment adherence.
Understanding of Treatment plan | 30 days.
  Assessing if the participant believes they have a good understanding of their care plan by self rating on a 7 point Likert Scale. Higher scores indicate greater understanding of treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Alana E Prejet, BScPN, BA, Principal Investigator — Brandon University
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No